CLINICAL TRIAL: NCT05193253
Title: Long-term Outcomes of Ablation, Liver Resection, and Liver Transplant as First-line Treatment for Solitary HCC of 3 cm or Less Using an Intention-to-treat Analysis: a Retrospective Cohort Study
Brief Title: Long-term Outcomes of Ablation, Liver Resection, and Liver Transplant as First-line Treatment for Solitary HCC of 3 cm or Less
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 16-5285.6
Record Dates: First submitted 2021-12-31; First posted 2022-01-14 (Actual); Last update posted 2022-01-18 (Actual); Status verified 2021-12

CONDITIONS: Hepatocellular Carcinoma
Keywords: liver transplant; liver resection; radiofrequency ablation; hepatocellular carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Radiofrequency Ablation; Hepatectomy; Liver Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Solitary HCC <= 3 cm: Treatment-naive patients with HCC <= 3 cm
  Interventions: Procedure: Radiofrequency ablation; Procedure: Liver resection; Procedure: Liver transplantation

INTERVENTIONS:
Procedure: Radiofrequency ablation — Treatment-naive patients with solitary HCC <= 3 cm who received ablation as the first-line treatment
Procedure: Liver resection — Treatment-naive patients with solitary HCC <= 3 cm who underwent liver resection as the first-line treatment
Procedure: Liver transplantation — Treatment-naive patients with solitary HCC <= 3 cm who were listed for liver transplantation as the first-line treatment

SUMMARY:
Curative-intent therapies for hepatocellular carcinoma (HCC) include radiofrequency ablation (RFA), liver resection (LR), and liver transplantation (LT). Controversy exists in treatment selection for early-stage tumors. We sought to evaluate the oncologic outcomes of patients who received either RFA, LR, or LT as first-line treatment for solitary HCC ≤ 3cm in an intention-to-treat analysis.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥18 years) patients
* Solitary HCC ≤ 3cm
* Receipt of either radiofrequency ablation, liver resection, or listing for a liver transplant
* Treatment received between Feb-2000 and Nov-2018

Exclusion Criteria:

* Pathology other than hepatocellular carcinoma (HCC)
* Receipt of prior treatment (i.e., not treatment naive)
* Not eligible for all of the three treatments (ablation, liver resection, or liver transplant listing)
* Platelet count <100,000 before treatment
* Alpha-1 fetoprotein (AFP) level > 1000 before treatment
* Age > 70 years
* Child-Pugh score C
* Esophageal varices grade greater than 2
* Model for End-stage Liver Disease (MELD) score before treatment exceeding 15
* Presence of ascites pretreatment
* Presence of encephalopathy pretreatment
* Spleen size greater than 12 cm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult (≥18 years) patients with solitary HCC ≤ 3cm who underwent either RFA, LR, or were listed for an LT between Feb-2000, and Nov-2018.
Sampling Method: Non-Probability Sample
Enrollment: 119 (Actual)
Dates: Start 2000-02-01 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2021-12-21 (Actual)

PRIMARY OUTCOMES:
Intention-to-treat (ITT) overall survival | Overall (median length of follow up of entire cohort 6.6 years)
  ITT was evaluated from the first treatment modality that was selected for curative intent. In the case of RFA and LR this was recorded as the time of the treatment. In the case of LT, the intention-to-treat was recorded at the time of listing for transplantation. The ITT analysis thus accounted for patients who were placed on the waitlist but dropped out.
Disease-free survival (DFS). | Overall (median length of follow up of entire cohort 6.6 years)
  DFS was defined as the time after treatment during which the patient was alive and free of disease. For DFS, patients were censored at recurrence, death, or loss to follow up.

IPD SHARING:
Plan to Share IPD: No
The data that support the findings of this study are unsuitable to post given that they contain potentially identifiable patient information. Moreover, the research ethics board at the University Health Network has only approved data to be stored and analyzed by the members of the institutional study team to minimize any breach of patient confidentiality.